CLINICAL TRIAL: NCT02498223
Title: Adjusting the Load Carried by the Soldier According to Body Composition Measurements and Aerobic Capacity
Acronym: LCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SHEBA-15-2156-OF-CTIL
Record Dates: First submitted 2015-06-17; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Work Load

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- research arm (Experimental): 50 subjects (healthy soldiers, male and female) from combat units will undergo the experiment protocol.
  Interventions: Other: experiment protocol

INTERVENTIONS:
Other: experiment protocol — the subjects will undergo the following experiment protocol:
  1. recruitment and medical examination day.
  2. physiological evaluation day- the subjects will perform twice* a physiological stress protocol ; 3 min sitting followed by 20 min walking on treadmill (4 km/h, 4% slope), and then 3 min sitting for recovery examination. total 26 min.
  3. biomechanical valuation day- the subjects will perform twice* a biomechanical protocol using the Zebris system; 2 min standing followed by 10 min walking on treadmill (4 km/h, 4% slope). total 12 min.
     * once carrying the weight calculated according to the army current instructions, and a second time carrying weight calculated according to the new LCI. 2 hours rest between the two performances.

SUMMARY:
In order to reduce the physiological and biomechanical loads that the soldiers are exposed to, the investigators want to examine new approaches for distributing the carried loads according to measurements that are specific for each soldier (body composition and aerobic capacity). A functional index (LCI=load carriage index) will provide the commander a tool for better decisions in distributing the same total load among the same number of soldiers, according to each soldier's ability.

DETAILED DESCRIPTION:
50 healthy, male and female combat soldiers will be recruited. Anthropometry and maximal aerobic capacity will be measured for each participant: Physiological evaluation: the participants will perform physical stress on a treadmill with changing slope and speed, once carrying 40% of their body weight (as the current instructions) and a second time with weight that is calculated by the examined body composition and aerobic capacity based index (LCI). The physiological response will be assessed based on heart rate, lactic acid in the blood and oxygen consumption.

Biomechanical evaluation: the biomechanical response will be measured in the biomechanical lab: pressure on the shoulder and waist from the load and straps, walk analysis and stress scatter in the foot.

By this experiment the investigators want to examine if the new index, the LCI, is physiologically and biomechanically better than the current load distribution instructions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-25 years.
* Healthy soldiers volunteers.
* Without heart, cardiovascular, metabolic or respiratory illnesses.
* Without known medical illness or medication use that might endanger the participants.

Exclusion Criteria:

* existence of any of undesired conditions detailed in the inclusion criteria.
* the physician decision.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-06 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
oxygen consumption | 3 experiment days
  oxygen consumption will be monitored continuously through the experimental days by a metabolic system (ERGOTEST 680, ZAN, GERMANY )

SECONDARY OUTCOMES:
Heart rate | 3 experiment days
  The heart rate will be monitored using a wearable heart rate monitor (Polar® sensor and heart rate monitor watch).
pressure at the shoulders and the waist | 3 experiment days
  pressure sensors will monitor the pressure from the load (carried on the back)
walk analysis (composite) | 3 experiment days
  analysing subject's walk using the Zebris Medical system. this system consist of a treadmill which is a FORCE PLATE that measure the forces between the treadmill and the shoe. the outcomes are diagram of vertical forces and walk pattern.

CONTACTS AND LOCATIONS:
Overall Officials: Ofir Frenkel, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Ramat- Gan, Israel